CLINICAL TRIAL: NCT07309029
Title: PROspective Evaluation of Pre-empTive Left Atrial Venoarterial Extra-Corporeal Membrane oxygenaTion for Complex High-risk Transcatheter Aortic Valve Replacement: PROTECT-TAVR
Brief Title: Pre-Emptive LAVA-ECMO for Complex High-Risk TAVR
Acronym: PROTECT-TAVR
Status: Recruiting | Type: Observational
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, Gennaro Giustino, MD, Atlantic Health System
Other Study IDs: 2337824
Record Dates: First submitted 2025-11-24; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Severe Aortic Stenosis; Cardiogenic Shock; Cardiogenic Shock, ECMO; Trans-catheter Aortic Valve Implantation
Keywords: severe aortic stenosis; cardiogenic shock; TAVR
MeSH Terms: conditions — Aortic Valve Stenosis; Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Left Atrial Veno-Arterial Extracorporeal Membrane Oxygenation (LAVA-ECMO) — Pre-emptive use of LAVA-ECMO involves transseptal cannulation of the left atrium to provide mechanical circulatory support and left ventricular unloading during high-risk transcatheter aortic valve replacement (TAVR). The device is placed prior to or at the start of the TAVR procedure in patients with unstable hemodynamics or complex anatomical features.

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility, effectiveness, and safety of pre-emptive left atrial veno-arterial extracorporeal membrane oxygenation (LAVA-ECMO) in patients undergoing complex and high-risk transcatheter aortic valve replacement (TAVR). These patients include adults with severe aortic stenosis who are hemodynamically unstable or at risk of instability due to anatomical complexity. The main questions it aims to answer are:

1. Does pre-emptive LAVA-ECMO reduce the incidence of in-hospital death, intraprocedural cardiac arrest, or emergent cardiac surgery?
2. What are the safety outcomes related to LAVA-ECMO, including major vascular, bleeding, or cardiac structural complications? -This is a single-arm, prospective, multi-center study with no comparison group.

Participants will:

* Be screened for eligibility based on hemodynamic status and anatomical complexity
* Undergo pre-emptive LAVA-ECMO cannulation prior to or during TAVR
* Receive follow-up assessments at 30 days and 1 year, including clinical evaluation and echocardiography

ELIGIBILITY:
Inclusion Criteria:

- Patients are required to have either a Class III hemodynamic status OR type B or type C anatomical complexity with Class II (at risk) hemodynamics (Figure 2).

* Hemodynamic Criteria

  * Major Criteria (Class III)

    * Systolic blood pressure <90 mmHg or MAP<60 mmHg
    * Need for vasopressors or inotropes to maintain MAP>60 mmHg
    * Evidence of end-organ damage including: acute kidney injury, liver dysfunction, elevated lactate or altered mentation
  * Minor Criteria (Class II)

    * Left ventricular ejection fraction <35%
    * Pulmonary hypertension (pulmonary artery systolic pressure >60 mmHg) with right ventricular dysfunction
    * Pulmonary capillary wedge pressure >30 mmHg
* Anatomic criteria

  * Major Criteria (Type C)

    * Native or valve-in-valve TAVR requiring single-leaflet modification for a large area of myocardium at risk (e.g. patients with large or dominant left circulation)
    * Native or valve-in-valve TAVR requiring dual-leaflet modification
    * Severe bioprosthetic aortic regurgitation
    * Severe 3-vessel coronary artery disease not amenable to revascularization (SYNTAX score >33)
  * Minor Criteria (Type B)

    * Native or valve-in-valve TAVR requiring single-leaflet modification
    * Severe commissural misalignment requiring leaflet modification
    * High-risk for coronary occlusion not amenable to leaflet modification
    * Critical low-flow low-gradient aortic stenosis (defined as an estimated aortic valve area ≤0.5 cm2)

Exclusion Criteria:

* Age <18 or pregnant

  * General absolute contraindications to TAVR
  * Severe peripheral artery disease with infeasibility for veno-arterial extracorporeal membrane oxygenation implantation.
  * Contraindications to transeptal cannulation (e.g. pre-existing interatrial septum occluder device).
  * Pre-existing Impella treatment.
  * Onset of shock >12 hours.
  * Preceding cardiac arrest with prolonged resuscitation (>40 minutes).
  * Other severe concomitant disease with life expectancy <6 months.
  * Participation in another trial with an intervention.
  * Any class I hemodynamic status
  * Type A anatomical complexity with class I or II hemodynamic status

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited from Atlantic Health System hospitals and affiliated centers. Eligible individuals are adult patients diagnosed with severe native aortic stenosis or degenerated bioprosthetic aortic valves who are scheduled for transcatheter aortic valve replacement (TAVR). Patients are identified through institutional clinical practices and referrals, including those admitted to the cardiac care unit with signs of hemodynamic instability or anatomical complexity. Recruitment may include critically ill patients who are sedated or intubated, with consent obtained from legally authorized representatives when necessary.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint: Composite of in-hospital death, intraprocedural resuscitated cardiac arrest or emergent cardiac surgery. | From enrollment through hospital discharge (up to 30 days post-procedure)

SECONDARY OUTCOMES:
Primary Safety Endpoint: Composite of VARC-3 major vascular complications, type 3 or 4 VARC-3 bleeding complications or major cardiac structural complications related to left atrial cannulation. | From enrollment through hospital discharge (up to 30 days post-procedure)
  The primary safety endpoint includes a composite of major vascular, bleeding and cardiac structural complications according to the VARC-3 criteria. For the purpose of this trial the component of the primary safety endpoint will be differentiated between TAVR-related (e.g. associated with the vascular access used for TAVR, valve delivery system or valve implant) and LAVA-ECMO-related (e.g. associated with LAVA-ECMO cannulation including transseptal puncture).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Center for Structural Heart Disease Henry Ford Hospital, Detroit, Michigan
  - Valve and Structural Heart Center Morristown Medical Center, Morristown, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] VARC-3 WRITING COMMITTEE:; Genereux P, Piazza N, Alu MC, Nazif T, Hahn RT, Pibarot P, Bax JJ, Leipsic JA, Blanke P, Blackstone EH, Finn MT, Kapadia S, Linke A, Mack MJ, Makkar R, Mehran R, Popma JJ, Reardon M, Rodes-Cabau J, Van Mieghem NM, Webb JG, Cohen DJ, Leon MB. Valve Academic Research Consortium 3: Updated Endpoint Definitions for Aortic Valve Clinical Research. J Am Coll Cardiol. 2021 Jun 1;77(21):2717-2746. doi: 10.1016/j.jacc.2021.02.038. Epub 2021 Apr 19. PMID 33888385
- [Background] Golzarian H, Thiel A, Hempfling G, Otto M, Otto T, Shappell E, Racer L, Martz D, Recker-Herman CM, Laird A, Cole WC, Sirak J, Patel SM. Severe aortic insufficiency-induced cardiogenic shock treated with left atrial VA-ECMO and emergent valve-in-valve TAVR. ESC Heart Fail. 2023 Dec;10(6):3718-3724. doi: 10.1002/ehf2.14561. Epub 2023 Oct 27. PMID 37890858
- [Background] Giustino G, O'Neill BP, Wang DD, Frisoli T, Fang JX, Engel-Gonzalez P, Lee J, Fadel R, O'Neill WW, Villablanca PA. Feasibility and safety of transcaval venoarterial extracorporeal membrane oxygenation in severe cardiogenic shock. EuroIntervention. 2024 Apr 15;20(8):e511-e513. doi: 10.4244/EIJ-D-23-01046. No abstract available. PMID 38629421
- [Background] Fraccaro C, Karam N, Mollmann H, Bleiziffer S, Bonaros N, Teles RC, Carrilho Ferreira P, Chieffo A, Czerny M, Donal E, Dudek D, Dumonteil N, Esposito G, Fournier S, Hassager C, Kim WK, Krychtiuk KA, Mehilli J, Pregowski J, Stefanini GG, Ternacle J, Thiele H, Thielmann M, Vincent F, von Bardeleben RS, Tarantini G. Transcatheter interventions for left-sided valvular heart disease complicated by cardiogenic shock: a consensus statement from the European Association of Percutaneous Cardiovascular Interventions (EAPCI) in collaboration with the Association for Acute Cardiovascular Care (ACVC) and the ESC Working Group on Cardiovascular Surgery. EuroIntervention. 2023 Oct 23;19(8):634-651. doi: 10.4244/EIJ-D-23-00473. PMID 37624587
- [Background] Villablanca PA, Al-Darzi W, Boshara A, Hana A, Basir M, O'Neill B, Frisoli T, Lee J, Wang DD, O'Neill WW. Left Atrial Venoarterial Extracorporeal Membrane Oxygenation for Patients in Cardiogenic Shock and Acute Aortic Regurgitation. JACC Cardiovasc Interv. 2022 Oct 24;15(20):2112-2114. doi: 10.1016/j.jcin.2022.08.015. Epub 2022 Sep 28. No abstract available. PMID 36265949
- [Background] Sabharwal A, Tsiouris A, Slaughter MS, Lemor A, Jeyakumar AKC, Protos A, Hernandez GA. Left Atrial-Veno Arterial Extracorporeal Membrane Oxygenation as a Bridge to Surgery for Endocarditis-Related Acute Severe Aortic Regurgitation. ASAIO J. 2024 Apr 1;70(4):e61-e64. doi: 10.1097/MAT.0000000000002077. Epub 2023 Nov 1. PMID 37913501
- [Background] Lemor A, Basir MB, O'Neill BP, Cowger J, Frisoli T, Lee JC, Wang DD, Alaswad K, O'Neill W, Villablanca PA. Left Atrial-Veno-Arterial Extracorporeal Membrane Oxygenation: Step-By-Step Procedure and Case Example. Struct Heart. 2022 Oct 31;6(6):100117. doi: 10.1016/j.shj.2022.100117. eCollection 2022 Nov. PMID 37288119
- [Background] Lama von Buchwald C, Gonzalez PE, O'Neill B, Wang DD, Frisoli T, O'Neill WW, Villablanca PA. Percutaneous Retrieval of an Aortic Valve Vegetation Causing Severe Regurgitation and Cardiogenic Shock. JACC Cardiovasc Interv. 2023 May 22;16(10):1301-1303. doi: 10.1016/j.jcin.2023.03.027. Epub 2023 May 3. No abstract available. PMID 37140503
- [Background] Fang JX, Giustino G, Apostolou D, Lee JC, Wang DD, Engel Gonzalez P, O'Neill BP, Frisoli TM, O'Neill WW, Villablanca PA. LAVA-ECMO-Supported Dual-Transcatheter Aortic and Mitral Valve-in-Valve Replacement in Cardiogenic Shock. JACC Case Rep. 2024 Oct 2;29(19):102564. doi: 10.1016/j.jaccas.2024.102564. eCollection 2024 Oct 2. PMID 39484326
- [Background] Chiang M, Gonzalez PE, O'Neill BP, Lee J, Frisoli T, Wang DD, O'Neill WW, Villablanca PA. Left Atrial Venoarterial Extracorporeal Membrane Oxygenation for Acute Aortic Regurgitation and Cardiogenic Shock. JACC Case Rep. 2022 Mar 2;4(5):276-279. doi: 10.1016/j.jaccas.2021.12.030. eCollection 2022 Mar 2. PMID 35257102
- [Background] Chiang M, Gonzalez PE, Basir MB, O'Neill BP, Lee J, Frisoli T, Wang DD, O'Neill WW, Villablanca PA. Modified Transcaval Left Atrial Venoarterial Extracorporeal Membrane Oxygenation Without Preplanning Contrast CT: Step-by-Step Guide. JACC Cardiovasc Interv. 2022 Aug 22;15(16):e181-e185. doi: 10.1016/j.jcin.2022.05.033. Epub 2022 Jul 13. No abstract available. PMID 35981853
- [Background] Nair RM, Chawla S, Alkhalaileh F, Abdelghaffar B, Bansal A, Higgins A, Lee R, Rampersad P, Khot UN, Jaber WA, Reed GW, Cremer PC, Menon V. Characteristics and Outcomes of Patients With Valvular Cardiogenic Shock. JACC Adv. 2024 Oct 4;3(11):101303. doi: 10.1016/j.jacadv.2024.101303. eCollection 2024 Nov. PMID 39429239
- [Background] Burkhoff D, Sayer G, Doshi D, Uriel N. Hemodynamics of Mechanical Circulatory Support. J Am Coll Cardiol. 2015 Dec 15;66(23):2663-2674. doi: 10.1016/j.jacc.2015.10.017. PMID 26670067
- [Background] Vincent JL, De Backer D. Circulatory shock. N Engl J Med. 2013 Oct 31;369(18):1726-34. doi: 10.1056/NEJMra1208943. No abstract available. PMID 24171518